CLINICAL TRIAL: NCT04322318
Title: Treatment of Newly Diagnosed Diffuse Anaplastic Wilms Tumors (DAWT) and Relapsed Favorable Histology Wilms Tumors (FHWT)
Brief Title: A Study of Combination Chemotherapy for Patients With Newly Diagnosed DAWT and Relapsed FHWT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AREN1921; NCI-2020-01561 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AREN1921 (Other: Children's Oncology Group); AREN1921 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2020-03-17; First posted 2020-03-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-04

CONDITIONS: Anaplastic Kidney Wilms Tumor; Recurrent Kidney Wilms Tumor; Stage II Kidney Wilms Tumor; Stage III Kidney Wilms Tumor; Stage IV Kidney Wilms Tumor
MeSH Terms: conditions — Wilms Tumor | interventions — Biopsy; Specimen Handling; Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Ifosfamide; Irinotecan; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; Surgical Procedures, Operative; Topotecan; Vincristine; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (Regimen UH-3) (Experimental): See outline in detailed description section.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Carboplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Procedure: Transabdominal Ultrasound; Drug: Vincristine; Procedure: X-Ray Imaging
- Arm II (Regimen ICE/Cyclo/Topo) (Experimental): CYCLES 1, 2, 4, 5, 7, AND 9: Patients receive carboplatin IV over 15-60 minutes on day 1. Patients also receive etoposide IV over 1-2 hours and ifosfamide IV over 2-4 hours on days 1-3. Treatment repeats every 21 days during cycles 1, 2, 4, 5, 7, and 9 in the absence of disease progression or unacceptable toxicity.
  CYCLES 3, 6, 8, AND 10: Patients receive cyclophosphamide IV over 15-30 minutes and topotecan IV over 30 minutes on days 1-5. Treatment repeats every 21 days during cycles 3, 6, 8, and 10 in the absence of disease progression or unacceptable toxicity.
  Patients undergo surgery and/or RT during cycles 4, 7, and 10 as clinically indicated. Patients undergo a CT scan, a PET scan, a chest x-ray, MRI, an abdominal ultrasound, and/or a bone scan throughout the trial. Patients may also undergo blood specimen collection and biopsy throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Carboplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Ifosfamide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Procedure: Surgical Procedure; Drug: Topotecan; Procedure: Transabdominal Ultrasound; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo a biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo a bone scan
  Other Names: Bone Scintigraphy
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
  Arms: Arm I (Regimen UH-3)
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
  Arms: Arm II (Regimen ICE/Cyclo/Topo)
Drug: Irinotecan — Given IV
  Arms: Arm I (Regimen UH-3)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo a PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Surgical Procedure — Undergo surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery
  Arms: Arm II (Regimen ICE/Cyclo/Topo)
Drug: Topotecan — Given IV
  Other Names: Hycamptamine; Topotecan Lactone
  Arms: Arm II (Regimen ICE/Cyclo/Topo)
Procedure: Transabdominal Ultrasound — Undergo abdominal ultrasound
  Other Names: abdominal ultrasound; TUS
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine
  Arms: Arm I (Regimen UH-3)
Procedure: X-Ray Imaging — Undergo a chest x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase II trial studies how well combination chemotherapy works in treating patients with newly diagnosed stage II-IV diffuse anaplastic Wilms tumors (DAWT) or favorable histology Wilms tumors (FHWT) that have come back (relapsed). Drugs used in chemotherapy regimens such as UH-3 (vincristine, doxorubicin, cyclophosphamide, carboplatin, etoposide, and irinotecan) and ICE/Cyclo/Topo (ifosfamide, carboplatin, etoposide, cyclophosphamide, and topotecan) work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. This trial may help doctors find out what effects, good and/or bad, regimen UH-3 has on patients with newly diagnosed DAWT and standard risk relapsed FHWT (those treated with only 2 drugs for the initial WT) and regimen ICE/Cyclo/Topo has on patients with high and very high risk relapsed FHWT (those treated with 3 or more drugs for the initial WT).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether the addition of vincristine/irinotecan to cyclophosphamide/ carboplatin/etoposide alternating with vincristine/doxorubicin/cyclophosphamide improves the event-free survival (EFS) of patients with newly diagnosed stage 4 diffuse anaplastic Wilms tumor (DAWT) as compared to historical controls.

II. To evaluate whether the addition of vincristine/irinotecan to cyclophosphamide/carboplatin/etoposide alternating with vincristine/doxorubicin/cyclophosphamide improves the EFS of patients with standard-risk relapsed favorable histology Wilms tumor (SRrFHWT) as compared to historical controls.

SECONDARY OBJECTIVES:

I. To evaluate whether the addition of vincristine/irinotecan to cyclophosphamide/carboplatin/etoposide alternating with vincristine/doxorubicin/cyclophosphamide improves the overall survival (OS) of patients with newly diagnosed stage 4 DAWT as compared to historical controls.

II. To evaluate whether the addition of vincristine/irinotecan to cyclophosphamide/carboplatin/etoposide alternating with vincristine/doxorubicin/cyclophosphamide improves the OS of patients with SRrFHWT as compared to historical controls.

III. To evaluate whether the addition of vincristine/irinotecan to cyclophosphamide/carboplatin/etoposide alternating with vincristine/doxorubicin/cyclophosphamide improves the EFS and OS of patients with newly diagnosed stage 2 and 3 DAWT as compared to historical controls.

IV. To establish EFS and OS for high-risk (HRrFHWT) and very high risk (VHRrFHWT) relapsed favorable histology Wilms tumor treated with ifosfamide/carboplatin/etoposide alternating with cyclophosphamide/ topotecan.

EXPLORATORY OBJECTIVES:

I. To describe renal toxicity of ifosfamide/carboplatin/etoposide in HRrFHWT and VHRrFHWT patients using conventional and novel biomarkers of renal toxicity (urine NGAL, cystatin C and Kim1) in the context of the chemotherapy regimens used on this study.

II. To collect and bank serial blood and urine samples in patients with newly diagnosed DAWT or relapsed FHWT and tumor tissue in patients with relapsed FHWT, for future analysis.

III. To assess the impact of p53 gene and protein expression on outcome for patients with newly diagnosed DAWT.

IV. To determine EFS/OS in the subsets of patients with newly diagnosed DAWT or relapsed FWHT who undergo gross total resection at all disease sites at diagnosis or after neoadjuvant chemotherapy.

V. To describe the rate of regional lymph node sampling at the time of nephrectomy with the use of a pre-operative surgical checklist for patients with newly diagnosed DAWT.

VI. To determine the feasibility of intensity modulated radiation therapy (IMRT) with central quality assurance (QA) monitoring to reduce radiation induced toxicity to the heart, thyroid, breast and solitary kidney for children with lung and liver metastases (part of an overarching aim in this study and across frontline favorable histology Wilms tumor studies).

VII. To validate that circulating tumor-derived deoxyribonucleic acid (ctDNA) can identify high-risk genomic features, define prognostic risk groups, and identify patterns of tumor evolution associated with the development of treatment resistance.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I (REGIMEN UH-3):

CYCLES 1, 5, 7, 10, AND 13: Patients receive vincristine intravenously (IV) via minibag per institutional policy on days 1, 8, and 15. Patients also receive doxorubicin IV over 1-15 minutes and cyclophosphamide IV over 30-60 minutes on day 1. Treatment repeats every 21 days during cycles 1, 5, 7, 10, and 13 in the absence of disease progression or unacceptable toxicity.

CYCLES 2, 6, 9, 12, AND 14: Patients receive carboplatin IV over 15-60 minutes on day 1. Patients also receive cyclophosphamide IV over 15-30 minutes and etoposide IV over 1-2 hours on days 1-4. Treatment repeats every 21 days during cycles 2, 6, 9, 12, and 14 in the absence of disease progression or unacceptable toxicity.

CYCLES 3, 4, 8, AND 11: Patients receive vincristine IV via minibag per institutional policy on days 1 and 8 and irinotecan IV over 90 minutes on days 1-5. Treatment repeats every 21 days during cycles 3, 4, 8, and 11 in the absence of disease progression or unacceptable toxicity.

Patients undergo radiation therapy (RT) at week 7 of cycle 3 as clinically indicated. Patients undergo a computed tomography (CT) scan, a positron emission tomography (PET) scan, a chest x-ray, magnetic resonance imaging (MRI), an abdominal ultrasound, and/or a bone scan throughout the trial. Patients may also undergo blood specimen collection and biopsy throughout the trial.

ARM II (REGIMEN IFOSFAMIDE, CARBOPLATIN, ETOPOSIDE [ICE]/CYCLOPHOSPHAMIDE [CYCLO]/TOPOTECAN [TOPO]):

CYCLES 1, 2, 4, 5, 7, AND 9: Patients receive carboplatin IV over 15-60 minutes on day 1. Patients also receive etoposide IV over 1-2 hours and ifosfamide IV over 2-4 hours on days 1-3. Treatment repeats every 21 days during cycles 1, 2, 4, 5, 7, and 9 in the absence of disease progression or unacceptable toxicity.

CYCLES 3, 6, 8, AND 10: Patients receive cyclophosphamide IV over 15-30 minutes and topotecan IV over 30 minutes on days 1-5. Treatment repeats every 21 days during cycles 3, 6, 8, and 10 in the absence of disease progression or unacceptable toxicity.

Patients undergo surgery and/or RT during cycles 4, 7, and 10 as clinically indicated. Patients undergo a CT scan, a PET scan, a chest x-ray, MRI, an abdominal ultrasound, and/or a bone scan throughout the trial. Patients may also undergo blood specimen collection and biopsy throughout the trial.

After completion of study treatment, patients are followed up every 3 months for years 1-2, every 6 months for years 3-4, and once at year 5.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed stages 2 - 4 diffuse anaplastic Wilms tumor must be enrolled on APEC14B1, consented to Part A - Eligibility Screening, and have received an initial stratum assignment showing DAWT (if anaplasia first identified at diagnostic, pre-treatment nephrectomy or biopsy) or a final stratum assignment showing DAWT (if anaplasia first noted at delayed nephrectomy) prior to enrollment on AREN1921. Prior enrollment on APEC14B1 is not an eligibility requirement for patients with relapsed favorable histology Wilms tumor.
* Patients must be =< 30 years old at study enrollment
* Patients with the following diagnoses are eligible for this study:

  * Newly diagnosed stages 2 - 4 diffuse anaplastic Wilms tumor as confirmed by central review
  * Favorable histology Wilms tumor at first relapse. Relapsed FHWT patients must have previously achieved remission for their initial FHWT diagnosis to be eligible for this study. The relapse risk groups are defined as follows, regardless of radiation therapy:

    * Standard-Risk relapse: Patients who received two chemotherapy agents for frontline therapy; primarily actinomycin D and vincristine
    * High-Risk relapse: Patients who received three chemotherapy agents for frontline therapy; primarily vincristine, actinomycin D and doxorubicin or vincristine, actinomycin D and irinotecan
    * Very High-Risk relapse: Patients who received four or more chemotherapy agents as part of initial therapy; primarily regimen M or its variations
* Patients with newly diagnosed DAWT must have had histologic verification of the malignancy. For relapsed FHWT patients, biopsy to prove recurrence is encouraged, but not required

  * Note: For relapsed FHWT patients, an institutional pathology report confirming favorable histology Wilms tumor (from relapse, if available, or from original diagnosis) must be available for upload prior to initiation of protocol therapy
* Patients with newly diagnosed Stages 2 - 4 diffuse anaplastic Wilms tumor must be enrolled on AREN1921 within 2 weeks of the tumor-directed surgery or biopsy procedure that first confirms a diagnosis of DAWT, whether at initial diagnostic procedure or delayed nephrectomy (such surgery/biopsy is day 0). For patients who received prior therapy for presumed favorable histology Wilms tumor, later confirmed to have diffuse anaplastic Wilms tumor at subsequent review of the initial biopsy
* Patients with newly diagnosed DAWT who undergo upfront nephrectomy must have at least 1 lymph node sampled prior to study enrollment
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients must have a life expectancy of >= 8 weeks
* Diffuse Anaplastic Wilms Tumor: Patients with diffuse anaplastic histology must have had no prior systemic therapy, except in the following situations:

  * Patients with diffuse anaplastic Wilms tumor who received no more than 12 weeks of pre nephrectomy chemotherapy for what was originally presumed to be favorable histology Wilms tumor, subsequently confirmed to be diffuse anaplastic Wilms tumor at delayed nephrectomy
  * Patients with diffuse anaplastic Wilms tumor who received no more than 6 weeks of chemotherapy following upfront biopsy, initiated within 14 days of biopsy, for presumed favorable histology Wilms tumor based on institutional review, but subsequently corrected to diffuse anaplastic Wilms tumor based on the initial stratum assignment on APEC14B1-REN
  * Treatment consisting of vincristine/doxorubicin/cyclophosphamide initiated on an emergent basis and within allowed timing as described
  * Note: Patients who received prior therapy for presumed favorable histology Wilms tumor, later identified to have diffuse anaplastic Wilms tumor as per above, must begin study treatment starting at cycle 3 (week 7) of regimen UH 3. Patients who received emergency radiation to preserve organ function are eligible as noted. Patients who received radiation as part of standard of care for presumed newly diagnosed favorable histology Wilms tumor, along with chemotherapy as noted above, prior to identification of diffuse anaplasia, are also eligible
* Relapsed Favorable Histology Wilms Tumor: Patients must not have received prior chemotherapy for their relapsed favorable histology Wilms tumor diagnosis. In addition, patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

  * Myelosuppressive chemotherapy: Must not have received within 2 weeks of entry onto this study
  * Radiation therapy (RT): >= 2 weeks (wks) must have elapsed for local palliative RT (small port); >= 6 months must have elapsed if prior craniospinal RT or if >= 50% radiation of pelvis; >= 6 wks must have elapsed if other substantial bone marrow (BM) radiation. Patients with relapsed favorable histology Wilms tumor who received emergency radiation to preserve organ function are eligible and do not need to washout with the above criteria
* Patients may not be receiving any other investigational agents (within 4 weeks prior to study enrollment)
* Peripheral absolute neutrophil count (ANC) >= 750/uL (performed within 7 days prior to enrollment)
* Platelet count >= 75,000/uL (transfusion independent) (performed within 7 days prior to enrollment)
* Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions) (performed within 7 days prior to enrollment)
* Patients with high-risk or very high-risk relapsed FHWT who will be treated with regimen ICE/Cyclo/Topo, must have renal function assessed by creatinine clearance or radioisotope glomerular filtration rate (GFR) and meet the following requirement:

  * Creatinine clearance or radioisotope GFR >= 60 mL/min/1.73 m^2 (performed within 7 days prior to enrollment)
* Patients diagnosed with stage 2-4 DAWT or standard risk relapsed FHWT, who will be treated with regimen UH 3, may either obtain a creatinine clearance, radioisotope GFR (meeting the above criteria of GFR >= 60 mL/min/1.73 m^2), or an adequate serum creatinine as per the following table:

  * Age: Maximum Serum Creatinine (mg/dL)
  * 1 month to < 6 months: 0.4 (male and female)
  * 6 months to < 1 year: 0.5 (male and female)
  * 1 to < 2 years: 0.6 (male and female)
  * 2 to < 6 years: 0.8 (male and female)
  * 6 to < 10 years: 1 (male and female)
  * 10 to < 13 years: 1.2 (male and female)
  * 13 to < 16 years: 1.5 (male), 1.4 (female)
  * >= 16 years: 1.7 (male), 1.4 (female)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age or direct bilirubin =< ULN for patients whose total bilirubin > 1.5 x ULN (performed within 7 days prior to enrollment)
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 x upper limit of normal (ULN) for age or =< 5 x ULN for patients with liver metastases (performed within 7 days prior to enrollment)
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by radionuclide angiogram (obtained within 21 days prior to enrollment and start of protocol therapy)

Exclusion Criteria:

* Patients with a history of bilateral Wilms tumor (synchronous or metachronous)
* Patients with any uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, or symptomatic congestive heart failure (defined as grade 2 or higher heart failure per Common Terminology Criteria for Adverse Events [CTCAE] version 5.0)
* Relapsed FHWT patients who did not receive frontline chemotherapy (e.g., very low risk FHWT initially observed without chemotherapy) or received only one chemotherapy agent for frontline therapy
* For patients with high-risk or very high-risk relapsed FHWT:

  * Patients with renal tubular acidosis (RTA) as evidenced by serum bicarbonate < 16 mmol/L and serum phosphate =< 2 mg/dL (or < 0.8 mmol/L) without supplementation
* For stages 2-4 DAWT and standard-risk relapsed FHWT patients:

  * Chronic inflammatory bowel disease and/or bowel obstruction
  * Concomitant use of St. John's wort, which cannot be stopped prior to the start of trial treatment
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 256 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) for stratum 1-3 | From study entry to the earliest of relapse or disease progression, second malignant neoplasm, or death from any cause, assessed up to 5 years from study entry
  Kaplan-Meier method will be used to estimate EFS, defined as the time from study entry until relapse or disease progression, secondary malignancy, or death.
EFS for stratum 4 | From study entry to the earliest of relapse or disease progression, second malignant neoplasm, or death from any cause, assessed up to 5 years from study entry
  Kaplan-Meier method will be used to estimate 4-year EFS, defined as the time from study entry until relapse or disease progression, secondary malignancy, or death.

SECONDARY OUTCOMES:
Overall survival (OS) for stratum 1-4 | From study entry to death due to any cause, assessed up to 5 years from study entry
  The Kaplan-Meier method will be used to estimate OS, defined as the time from study entry until death.

OTHER OUTCOMES:
Percentage of patients experiencing grade 3+ renal adverse events | Up to 30 weeks on average for Stratum 4 only
  Percentage of patients experiencing grade 3 or higher renal adverse events. Will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Collection of blood and urine samples | Up to 42 weeks on average for Strata 1-3 and up to 30 weeks on average for Stratum 4
  For all Strata 1-4, serial blood and urine samples will be collected (during protocol therapy, at the end of protocol therapy, and at first relapse) and banked for future analysis such as evaluation of minimal residual disease by assessing levels of circulating tumor-derived deoxyribonucleic acid (ctDNA).
p53 biomarker analysis | Based on tissue collected at diagnosis (Strata 1 and 2 only), with outcomes collected up to 5 years after study entry
  For patients with diffuse anaplastic Wilms tumors (DAWT) (Strata 1 and 2), p53 from diagnostic tissue will be assessed, and rates of p53 mutations described overall and within each stratum. Degree of anaplasia as a predictor of p53 mutation status will be analyzed in logistic regression models, and association of p53 status with EFS and OS will be analyzed in Cox regression models, stratified by disease stage. Possible interactions between p53 mutation status and degree of anaplasia in outcome models will be explored.
EFS for patients with gross total disease resection | Up to 5 years after study entry
  EFS will be described for newly diagnosed disease stage 2-4 DAWT patients (Strata 1 and 2) and relapsed favorable histology Wilms tumors (FHWT) patients (Strata 3 and 4) who have gross total disease resection prior to enrollment or at the time of delayed nephrectomy following adjuvant chemotherapy. Kaplan-Meier curves will be reported by strata with 95% confidence bands. Potential prognostic factors for these patients will be explored in Cox regression models.
OS for patients with gross total disease resection | Up to 5 years after study entry
  OS will be described for newly diagnosed disease stage 2-4 DAWT patients (Strata 1 and 2) and relapsed FHWT patients (Strata 3 and 4) who have gross total disease resection prior to enrollment or at the time of delayed nephrectomy following adjuvant chemotherapy. Kaplan-Meier curves will be reported by strata with 95% confidence bands. Potential prognostic factors for these patients will be explored in Cox regression models.
Association of the number of nodes examined with EFS and OS | Nodal information from upfront or delayed nephrectomy, with outcomes collected for up to 5 years after study entry
  The number of lymph nodes examined at the time of primary nephrectomy and number of positive nodes will be collected for all DAWT patients who enroll to Strata 1 or 2. The association of the number of nodes examined with EFS and OS will be explored in Cox regression models stratified by disease stage. For each of these analyses, association will be expressed either as a single hazard ratio if the effect is found to be linear, or as continuous functions on the hazard ratio scale if the effect is found to be non-linear. Similar models will be fit to examine the association between ratio of positive nodes to nodes examined and outcomes. Confidence intervals or bands will be reported for all quantities.
Rates of usage of intensity-modulated radiation therapy | Up to 7 or 30 weeks
  Will be reported descriptively for cohorts receiving radiation.
Detection and quantification of ctDNA | Up to 42 weeks on average for Strata 1-3 and up to 30 weeks on average for Stratum 4
  Presence/absence of ctDNA at study entry (diagnosis for DAWT Strata 1 and 2, and first relapse for relapsed FHWT Strata 3 and 4) as well as ctDNA levels as a continuous variable will be associated with subsequent EFS using Kaplan-Meier methodology, log-rank tests, and Cox proportional hazards modeling. ctDNA over time (diagnosis, on treatment, and off treatment) will be associated with clinical outcomes using longitudinal modeling. Where sufficient EFS events exist, ctDNA will be evaluated alongside or in combination with other known risk factors to establish risk groups. Genomic features such as TP53 and 1q gain identified in ctDNA will be reported descriptively and correlated with tumor-based marker findings.

CONTACTS AND LOCATIONS:
Overall Officials: James I Geller, Principal Investigator — Children's Oncology Group
Locations (204):
- United States (177):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Monash Medical Center-Clayton Campus, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (14):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (2):
  - HIMA San Pablo Oncologic Hospital, Caguas
  - University Pediatric Hospital, San Juan
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia